CLINICAL TRIAL: NCT00263471
Title: Phase 2 Study of the Effect of 7-Methylxanthine on the Progression of Childhood Myopia
Brief Title: Myopia Progression and the Effect of 7-Methylxanthine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Trier Research Laboratories (Other)
Collaborators: Generalkonsul Einar Høyvalds Fond (Unknown); Jørgen Bagenkop Nielsens Myopi-Fond (Unknown); Chr. Andersen og hustru Ingeborg Andersen, f. Schmidts legat (fond) oprettet af deres datter, frk. Lilli Ellen Andersen. (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2612-2320
Record Dates: First submitted 2005-12-06; First posted 2005-12-08 (Estimated); Last update posted 2005-12-14 (Estimated); Status verified 2003-10

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — 7-methylxanthine

INTERVENTIONS:
Drug: 7-methylxanthine

SUMMARY:
7-methylxanthine has been shown to increase the concentration and thickness of collagen fibrils in rabbit sclera. Deficient collagen in the sclera may be the cause of progression of childhood myopia. The study hypothesis is that treatment with 7-methylxanthine will stabilize the sclera and prevent further progression of myopia.

DETAILED DESCRIPTION:
Participants are given tablets of 7-methylxanthine 400 mg per day or placebo tablets for 12 months. Axial length, cycloplegic refraction and corneal curvature is measured, as well as weight, height, blood pressure and heart rate. The participants are interviewed about possible CNS, gastrointestinal, or cardiopulmonal side effects.

ELIGIBILITY:
Inclusion Criteria:

Children in the age 8-13 years with myopia and an axial growth rate of 0.15 mm or more per year.

-

Exclusion Criteria:

Severe general ailment (for example diabetes, epilepsy, psychiatric disease) Eye diseases (for example cataract, keratoconus, chronic iritis, glaucoma)

-

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90
Dates: Start 2003-10; Study Completion 2006-03

PRIMARY OUTCOMES:
Axial growth

SECONDARY OUTCOMES:
Myopia progression

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Trier, MD, Study Chair — Trier Research Laboratories

REFERENCES:
- [Background] Trier K, Olsen EB, Kobayashi T, Ribel-Madsen SM. Biochemical and ultrastructural changes in rabbit sclera after treatment with 7-methylxanthine, theobromine, acetazolamide, or L-ornithine. Br J Ophthalmol. 1999 Dec;83(12):1370-5. doi: 10.1136/bjo.83.12.1370. PMID 10574816
- [Derived] Lawrenson JG, Shah R, Huntjens B, Downie LE, Virgili G, Dhakal R, Verkicharla PK, Li D, Mavi S, Kernohan A, Li T, Walline JJ. Interventions for myopia control in children: a living systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 16;2(2):CD014758. doi: 10.1002/14651858.CD014758.pub2. PMID 36809645
- [Derived] Cui D, Trier K, Munk Ribel-Madsen S. Effect of day length on eye growth, myopia progression, and change of corneal power in myopic children. Ophthalmology. 2013 May;120(5):1074-9. doi: 10.1016/j.ophtha.2012.10.022. Epub 2013 Feb 4. PMID 23380471